CLINICAL TRIAL: NCT03656315
Title: Proposal for a Scoring System to Predict the Depth of Cricothyroid Membrane by Correlating Airway Assessment Parameters to the Depth of Cricothyroid Membrane
Brief Title: Scoring System to Predict Depth of Cricothyroid Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Principal Investigator, Cyprican Mendonca, Consultant Anaesthetist, University Hospitals Coventry and Warwickshire NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 247781
Record Dates: First submitted 2018-08-15; First posted 2018-09-04 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2021-03

CONDITIONS: Airway Obstruction
Keywords: Difficult airway; Cricothyroid membrane; Assessment
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Intervention Model Description: All recruited participants will be included in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Airway assessment (Other): All patients recruited will be entered into this arm of the study. Airway assessment including Ultrasound scan will be performed
  Interventions: Other: Airway Assessment

INTERVENTIONS:
Other: Airway Assessment — All patients recruited to this study will have an ultrasound of their cricothyroid membrane

SUMMARY:
This study looks to devise a scoring system that can be used to predict difficult front of neck access due to increased depth of cricothyroid membrane. This study will recruit elective patients undergoing operations for a variety of procedures and correlate their measured (by ultrasound) cricothyroid depth with other difficult airway predictors (such as Mallampatti score).

DETAILED DESCRIPTION:
A 'can't intubate can't oxygenate scenario (CICO) is defined as a situation when there is a failed intubation and failure to adequately oxygenate using facemask ventilation or supraglottic airway device resulting in increasing hypoxemia in an anaesthetised and paralysed patient. Although this situation is rare, if not managed appropriately it can result in hypoxic brain damage and death. The successful management of CICO includes timely decision making to perform front of neck access (FONA) via the cricothyroid membrane (CTM). The currently recommended technique in the UK is surgical cricothyroidotomy.

Successful FONA depends on the ease of anatomy of the neck and the ability to locate the cricothyroid membrane. In cases where the cricothyroid membrane is not palpable, front of neck access is difficult. The clinical procedure involves an 8 cm long skin incision and finger dissection to palpate the cricothyroid membrane. In a real-life situation, this will be compounded by profuse bleeding and no structure would be visible. Therefore, prediction of difficult FONA and appropriate preparation is essential for safe airway management.

Routine airway assessment includes mouth opening measured as inter-incisor gap, Mallampatti score, thyromental distance, sternomental distance, jaw protrusion and neck movements. In addition, ability to perform front of neck access should be ascertained prior to induction of general anaesthesia. Depth of cricothyroid membrane is one of the factors leading to technical difficulties in front of neck access. In situations where the CTM is deep and not palpable, FONA is technically difficult and takes longer. A previous observational study has shown a positive correlation between patient's weight, height, body mass index and neck circumference with depth of cricothyroid membrane. A scoring system to assess the depth of cricothyroid membrane based on the patient's height, weight, neck circumference and other airway assessment parameters would be useful in predicting the depth of CTM. Hence difficulties with front of neck access can be anticipated and appropriate measures can be taken in the event a CICO situation arises.

DAS 2015 guideline recommend airway assessment and preparation for all patients presenting for surgery. Routine airway assessment includes mouth opening measured as inter-incisor gap, Mallampatti score, thyromental distance, sternomental distance, jaw protrusion and neck movements. In addition, ability to perform front of neck access should be ascertained prior to induction of general anaesthesia. Depth of cricothyroid membrane is one of the factors leading to technical difficulties in front of neck access. In situations where the CTM is deep and not palpable, FONA is technically difficult and takes longer. A previous observational study has shown a positive correlation between patient's weight, height, body mass index and neck circumference with depth of cricothyroid membrane. A scoring system to assess the depth of cricothyroid membrane based on the patient's height, weight, neck circumference and other airway assessment parameters would be useful in predicting the depth of CTM. Hence difficulties with front of neck access can be anticipated and appropriate measures can be taken in the event a CICO situation arises.

ELIGIBILITY:
Inclusion Criteria:

* Elective cases

Exclusion Criteria:

* Emergency cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Correlation between difficult airway indicators and cricothyroid membrane | 20 minutes
  A positive correlation between airway assessment parameters and depth of the cricothyroid membrane

SECONDARY OUTCOMES:
A scoring system to predict the depth of cricotyroid membrane | 20 minutes
  A scoring system to predict the depth of the cricothyroid membrane using airway assessment parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom